CLINICAL TRIAL: NCT06209814
Title: Evaluation of Open-face Maxillary Complete Denture for Patients With Prominent Premaxilla. Crossover Study
Brief Title: Evaluation of Open-face Maxillary Complete Denture for Patients With Prominent Premaxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: haitham ahmed hassan ismail (Other)
Responsible Party: Sponsor-Investigator, haitham ahmed hassan ismail, Assistant Lecturer of Prosthodontics, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0672-04/2023
Record Dates: First submitted 2024-01-06; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Edentulous Jaw
Keywords: Prominent Premaxilla
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional denture (Active Comparator)
  Interventions: Device: Conventional denture
- maxillary open-faced denture (Experimental)
  Interventions: Device: Maxillary open-faced denture

INTERVENTIONS:
Device: Conventional denture — Patients in this group received conventional maxillary and mandibular complete dentures. The patients used these dentures for 45 days. Then, the conventional maxillary denture was replaced by open faced denture with soft acryl resin wing.
  Arms: Conventional denture
Device: Maxillary open-faced denture — Patients in this group received a maxillary open faced denture with soft acryl resin wing and a conventional mandibular complete denture. The patients used these dentures for 45 days. Afterward, the maxillary open-faced denture was replaced by one with a conventional construction.
  Arms: maxillary open-faced denture

SUMMARY:
The aim of the present study was to evaluate open faced maxillary complete denture with soft acryl resin wing versus conventional heat cured maxillary complete denture regarding the retention and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous male patients.
* Patients having had no previous complete dentures
* Patients with well-developed edentulous ridge with proclined premaxilla covered with healthy firm mucosa
* Patients with normal Angle Class 1 maxillomandibular relationship

Exclusion Criteria:

* Patients with resorbed ridges
* Patients with xerostomia and patients undertaking medications that affect salivary flow (e.g., diuretics). Similarly, patients with systemic diseases that may affect the amount or consistency of saliva (e.g., uncontrolled diabetes mellitus).

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Denture retention | up to 45 days
  Evaluated using a universal testing machine to exert a vertical dislodging force on the denture. A stainless-steel loop was attached to the geometric center of the denture using autopolymerizing acrylic resin. The center of the labial frenum (point A) and the hamular notches (points B&C) were located in the denture base. The distance halfway between points B and C was measured, and the location was marked on the posterior border of the denture base (point D). Half the distance between points A and D was marked as the denture base center (point E). A force transmission device was used to transmit the dislodging vertical force from the universal testing machine to the denture. A facebow was used to set the Frankfort plane of the patient parallel to the floor. After orienting the participant to the testing machine, it was set to exert a dislodging force at a rate of 50 mm/min. The test was repeated 3 times for each denture and the mean was calculated.
Patient satisfaction with esthetics | up to 45 days
  Participant satisfaction with esthetics was evaluated by using a Visual Analogue Scale (VAS). The level of satisfaction was indicated as a sign on a 10 cm VAS, labeled with (not at all satisfied) at the zero end with (completely satisfied) at the other end. The distance (mm) between the zero point and the sign marked by the patient on the 10-cm-line was measured and expressed in percentage.
Patient satisfaction with comfort | up to 45 days
  Participant satisfaction with comfort was evaluated by using a Visual Analogue Scale (VAS). The level of satisfaction was indicated as a sign on a 10 cm VAS, labeled with (not at all satisfied) at the zero end with (completely satisfied) at the other end. The distance (mm) between the zero point and the sign marked by the patient on the 10-cm-line was measured and expressed in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Haitham A Ismail, MSc, Principal Investigator — Alexandria University; Ingy S Soliman, PhD, Study Chair — Alexandria University; Muhammed B El-Danasory, PhD, Study Chair — Alexandria University; Salma S Abolgheit, PhD, Study Chair — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt